CLINICAL TRIAL: NCT01045707
Title: NN5401-3590: A Trial Comparing Efficacy and Safety of NN5401 With Insulin Glargine in Insulin Naive Subjects With Type 2 Diabetes (BOOST™ : START 1) / NN5401-3726: An Extension Trial Comparing Safety and Efficacy of NN5401 With Insulin Glargine in Subjects With Type 2 Diabetes (BOOST™: START 1)
Brief Title: Comparison of NN5401 Versus Insulin Glargine, Both Combined With Metformin Treatment, in Subjects With Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3590; 2009-011271-78 (EudraCT Number); U1111-1111-7178 (Other: WHO); 2009-015839-33 (EudraCT Number); U1111-1114-9237 (Other: WHO); NCT01169766 (obsolete NCT alias)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp OD (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IGlar OD (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected s.c. (under the skin) once daily with the breakfast meal. Dose was individually adjusted.
  Arms: IDegAsp OD
Drug: insulin glargine — Injected s.c. (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of this trial is to compare the efficacy and safety of NN5401 (insulin degludec/insulin aspart (IDegAsp)) with insulin glargine (IGlar), both as add-on to subject's ongoing treatment with metformin + at least one OAD (oral anti-diabetic drug).

The main period is registered internally at Novo Nordisk as NN5401-3590 while the extension period is registered as NN5401-3726.

ELIGIBILITY:
Inclusion Criteria:

* For MAIN period (NN5401-3590):
* Diagnosis of type 2 diabetes mellitus for at least 6 months
* Insulin naïve subjects
* Treatment with metformin and at least one other oral antidiabetic drug for at least 3 months before trial start
* Glycosylated haemoglobin (HbA1c) between 7.5 - 11.0% (both inclusive)
* Body Mass Index (BMI) no higher than 40.0 kg/m^2
* For EXTENSION period (NN5401-3726):
* Informed consent obtained before any trial-related activities
* Must have completed the 26-week treatment period (visit 28) in trial NN5401-3590

Exclusion Criteria:

* For MAIN period (NN5401-3590):
* Treatment with glucagon like peptide-1 (GLP-1) receptor agonists and/or thiazolidinedione(s) within the last 3 months prior to trial start
* Cardiovascular disease diagnosed within 6 months before trial start
* For EXTENSION period (NN5401-3726):
* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as systemic corticosteroids, beta-blockers, Monoamine oxidase (MAO) inhibitors
* Anticipated significant lifestyle changes during the trial, e.g. shift work (including permanent night/evening shift workers), as well as highly variable eating habits as judged by the physician)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (78):
- United States (36):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, North Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Springfield, Missouri
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Wilson, North Carolina
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Tomball, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
- Austria (5):
  - Novo Nordisk Investigational Site, Ebreichsdorf
  - Novo Nordisk Investigational Site, Feldbach
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- India (6):
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Trichy, Tamil Nadu
  - Novo Nordisk Investigational Site, Bangalore
  - Novo Nordisk Investigational Site, Kerala
  - Novo Nordisk Investigational Site, Patna
- Poland (5):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Pruszków
  - Novo Nordisk Investigational Site, Warsaw
- Novo Nordisk Investigational Site, Bayamón, Puerto Rico
- Russia (9):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Orenburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Yaroslavl
- South Korea (3):
  - Novo Nordisk Investigational Site, Pucheon
  - Novo Nordisk Investigational Site, Pusan
  - Novo Nordisk Investigational Site, Seoul
- Spain (11):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Mérida
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Partida de Bacarot
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, San Sebastián de los Reyes
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Kumar A, Franek E, Wise J, Niemeyer M, Mersebach H, Simo R. Efficacy and Safety of Once-Daily Insulin Degludec/Insulin Aspart versus Insulin Glargine (U100) for 52 Weeks in Insulin-Naive Patients with Type 2 Diabetes: A Randomized Controlled Trial. PLoS One. 2016 Oct 19;11(10):e0163350. doi: 10.1371/journal.pone.0163350. eCollection 2016. PMID 27760129
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 88 sites in 8 countries: Austria (4), India (7), South Korea (5), Poland (6), Russia (10), Spain (11), Turkey (5), and United States of America (40). Some sites did not enroll subjects in the extension period.
Pre-assignment Details: The total duration of treatment was up to 52 weeks (26 weeks [main trial: NN5401-3590, NCT01045707] + 26 weeks [extension trial: NN5401-3726]), separated by 1 week of wash-out period; during which subjects were treated with Neutral Protamine Hagedorn (NPH) insulin twice daily (BID) in combination with subject's pre-trial treatment of metformin.
Groups:
- IDegAsp OD: Insulin degludec/insulin aspart (IDegAsp) was given subcutaneously (s.c.) once daily (OD) in combination with subject's pre-trial treatment of metformin. IDegAsp was given with breakfast for 26 weeks in the main period and with either breakfast or with the largest meal for another 26 weeks in the extension period.
- IGlar OD: Insulin glargine (IGlar) was given subcutaneously (s.c.) once daily (OD) according to approved labelling in combination with subject's pre-trial treatment of metformin. IGlar was given for 52 weeks (26 weeks in main period and 26 weeks in extension period).
Period: Main: Week 0 to 26 (NN5401-3590)
Arm/Group | IDegAsp OD | IGlar OD
Started | 266 | 264
Exposed | 265 (One subject withdrew prior to exposure to trial drug) | 261 (Three subjects withdrew prior to exposure to trial drug)
Completed | 219 | 232
Not Completed | 47 | 32
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 4 | 2
Not completed — Protocol Violation | 6 | 5
Not completed — Withdrawal Criteria | 22 | 11
Not completed — Unclassified | 10 | 11
Period: Extension: Week 27 to 52 (NN5401-3726)
Arm/Group | IDegAsp OD | IGlar OD
Started | 192 (Twenty seven subjects from main trial did not continue into the extension) | 221 (Eleven subjects from main trial did not continue into the extension)
Completed | 179 | 209
Not Completed | 13 | 12
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal criteria | 2 | 1
Not completed — Unclassified | 6 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for all the randomised subjects (the full analysis set [FAS]) were collected at the beginning of main trial. One subject was excluded from FAS because the subject was randomised in error and was not dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp OD | IGlar OD | Total
Number analyzed (Participants) | 266 | 263 | 529
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.0) | 56.4 (9.2) | 56.9 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 141 | 127 | 268
  Male | 125 | 136 | 261
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.9 (1.0) | 8.9 (0.9) | 8.9 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.1 (2.9) | 10.4 (2.8) | 10.2 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). One subject was excluded from FAS because the subject was randomised in error and was not dosed.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 266 | 263
percentage of glycosylated haemoglobin | -1.65 (1.28) | -1.72 (1.17)

2. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment.
Time Frame: Week 0, Week 53
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 266 | 263
percentage of glycosylated haemoglobin | -1.39 (1.23) | -1.34 (1.16)

3. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 26
Description: Mean of SMPG at 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). One subject was excluded from FAS because the subject was randomised in error and was not dosed. For 24 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 256 | 249
mmol/L | 7.9 (2.1) | 7.9 (1.7)

4. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 53 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 265 | 261
Episodes/100 years of patient exposure | 419 | 211

5. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 53 + 7 days follow up
Population: as for outcome 4
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 265 | 261
Episodes/100 years of patient exposure | 19 | 53

6. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild:no or transient symptoms, no interference with the subject's daily activities. Moderate: marked symptoms, moderate interference with the subject's daily activities. Severe: considerable interference with the subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalisation/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect
Time Frame: Week 0 to Week 53 + 7 days follow up
Population: as for outcome 4
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 265 | 261
Events/100 years of patient exposure
  Adverse events (AE) | 313 | 238
  Serious AE | 17 | 9
  Severe AE | 9 | 10
  Moderate AE | 77 | 66
  Mild AE | 227 | 162
  Fatal AE | 2 | 1

ADVERSE EVENTS:
Time Frame: Week 0 to Week 53 + 7 days follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 30/265 | 15/261
Other Adverse Events (participants affected / at risk) | 88/265 | 79/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=265) | IGlar OD (N=261)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=265) | IGlar OD (N=261)
Nasopharyngitis (Infections and infestations) | 36 (47) | 35 (51)
Headache (Nervous system disorders) | 16 (19) | 11 (20)
Hypertension (Vascular disorders) | 20 (23) | 11 (12)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (24) | 11 (15)
Upper Respiratory Tract Infection (Infections and infestations) | 15 (17) | 12 (18)
Bronchitis (Infections and infestations) | 14 (15) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 13 (20) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.